CLINICAL TRIAL: NCT01344200
Title: CELECOXIB Plasma and Cerebral Spinal Fluid Pharmacokinetics in Children
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Hospital of Eastern Ontario (Other)
Responsible Party: Principal Investigator, Kimmo Murto, Director of Research, Department of Anesthesiology & Pain Medicine, Children's Hospital of Eastern Ontario
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 09/09E
Record Dates: First submitted 2011-04-21; First posted 2011-04-29 (Estimated); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Pharmacokinetics of Celecoxib in Children
Keywords: Pharmacokinetics; Celecoxib; Children; Pharmacogenetic; ABCB1 genotype; CYP2C9 genotype; CSF; Plasma
MeSH Terms: interventions — Celecoxib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Phase I: Study drug Group 1 (Celecoxib 7 mg/kg) (Active Comparator): Study participants randomized to this group will receive a single 7 mg/kg dose of celecoxib approximately 121-180 minutes before their scheduled LP ± BMA. The study medication will be a liquid and the study participant will be asked to drink it.
  Interventions: Drug: Celecoxib
- Phase I: Study drug Group 2 (Celecoxib 14 mg/kg) (Active Comparator): Study participants randomized to this group will receive a single 14 mg/kg dose of celecoxib approximately 121-180 minutes before their scheduled LP ± BMA. The study medication will be a liquid and the study participant will be asked to drink it.
  Interventions: Drug: Celecoxib
- Phase II: Group A: Placebo (Placebo Comparator): Study participants will receive a single dose of placebo. Placebo will be liquid. The study participant will drink it.
  The timing of when the study participants in this group will take placebo will be determined in a second randomization:
  Group A.1: will take placebo 15 to 24 hours prior to having their LP±BMA. The study medication will be taken at home.
  Group A.2: will take placebo 5 to 15 hours prior to having their LP±BMA. The study medication will be taken at home.
  Group A.3: will take the placebo 3 to 5 hours prior to having their LP±BMA. The study medication will be taken at home.
  Group A.4: will take the study medication 1 to 2 hours prior to having their LP±BMA. The study medication will be taken at the hospital.
  Group A.5: will take the study medication 0 to 60 minutes prior to having their LP±BMA. The study medication will be taken at the hospital.
  Interventions: Drug: Placebo
- Phase II: Group B: Study drug (Celecoxib 7 mg/kg) (Active Comparator): Study participants randomized to this group you will receive a single 7 mg/kg dose of celecoxib which will be in a liquid form, and the study participant will drink it.
  The timing of when the study participant in this group will take this medication will be determined in a second randomization:
  Group B.1: will take the study medication 15 to 24 hours prior to having their LP±BMA. The study medication will be taken at home.
  Group B.2: will take the study medication 5 to 15 hours prior to having their LP±BMA. The study medication will be taken at home.
  Group B.3: will take the study medication 3 to 5 hours prior to having their LP±BMA. The study medication will be taken at home.
  Group B.4: will take the study medication 1 to 2 hours prior to having their LP±BMA. The study medication will be taken at the hospital.
  Group B.5: will take the study medication 0 to 60 minutes prior to having your LP±BMA. The study medication will be taken at the hospital.
  Interventions: Drug: Celecoxib
- Phase II: Group C: Study drug (Celecoxib 14 mg/kg) (Active Comparator): Study participants randomized to this group you will receive a single 14 mg/kg dose of celecoxib which will be in a liquid form, and the study participant will drink it.
  The timing of when the study participant in this group will take this medication will be determined in a second randomization:
  Group C.1: will take the study medication 15 to 24 hours prior to having their LP±BMA. The study medication will be taken at home.
  Group C.2: will take the study medication 5 to 15 hours prior to having their LP±BMA. The study medication will be taken at home.
  Group C.3: will take the study medication 3 to 5 hours prior to having their LP±BMA. The study medication will be taken at home.
  Group C.4: will take the study medication 1 to 2 hours prior to having your LP±BMA. The study medication will be taken at the hospital.
  Group C.5: will take the study medication 0 to 60 minutes prior to having your LP±BMA. The study medication will be taken at the hospital.
  Interventions: Drug: Celecoxib

INTERVENTIONS:
Drug: Celecoxib — In Phase I twenty (20) children will receive either celecoxib 14 or 7 mg/kg 120-180 minutes prior to lumbar puncture (LP). In Phase II forty-five (45) children will receive celecoxib 14 mg/kg, 7 mg/kg or placebo in one of 5 time intervals, 1-24 hours prior to LP.
  Other Names: Celebrex
  Arms: Phase I: Study drug Group 1 (Celecoxib 7 mg/kg); Phase I: Study drug Group 2 (Celecoxib 14 mg/kg); Phase II: Group B: Study drug (Celecoxib 7 mg/kg); Phase II: Group C: Study drug (Celecoxib 14 mg/kg)
Drug: Placebo — In Phase II forty-five (45) children will receive celecoxib 14 mg/kg, 7 mg/kg or placebo in one of 5 time intervals, 1-24 hours prior to LP.
  Arms: Phase II: Group A: Placebo

SUMMARY:
Celecoxib is effective for reducing postoperative pain in adults. Children use celecoxib more rapidly than adults and require higher doses. Celecoxib is partially metabolized in the liver by a certain enzyme. A person's genetic variation of this enzyme can influence how well their body uses Celecoxib. Furthermore, Celecoxib down-regulates P-glycoprotein (P-gp), a drug efflux transporter located at the blood brain barrier responsible for central nervous system (CNS) extrusion of ondansetron and possibly fentanyl; therefore celecoxib may augment the CNS effects of these drugs.

Understanding the blood and cerebrospinal fluid (CSF) profile of celecoxib in children and the influence of genetics on metabolism would help to develop appropriate celecoxib dosing in children for various treatment options.

DETAILED DESCRIPTION:
Background:

Celecoxib is a selective cyclooxygenase-2 (Cox-2) inhibitor belonging to the non-steroidal anti-inflammatory drugs (NSAIDs) class of medications. Adult studies have evaluated single dose and short term courses of Celecoxib and shown improved postoperative analgesia. One pharmacokinetic (PK) study suggested that celecoxib had faster clearance in pediatric patients implying the need for a higher dose in children. Adult literature has reported Cox-2 inhibitor administration up to 10 times the typical dose without adverse side effects. One adult chemotherapy drug trial involved high dose Celecoxib for a median of 8.4 months with very limited side effects. Another study demonstrated that blood brain barrier (BBB) permeable selective Cox-2 inhibitors effectively reduced central nervous system Prostaglandin (PG) E2, (a surrogate marker of Cox-2 activity) concentrations and postoperative pain.

Celecoxib may influence CSF levels of various drugs, possibly via a P-gp regulation mechanism. Brain uptake of drugs is limited by both an anatomic (passive) and a biochemical (active) blood brain barrier (BBB). Metabolic enzymes and efflux protein transport systems represent the latter; the best known group is the ATP-binding cassette (ABC) protein transporters and best studied is P-gp encoded by the ABCB1 (aka MDR1) gene. P-gp actively pumps drugs and toxins out of the central nervous system (CNS) and acts in concert with detoxification enzymes to defend against cell damage. Celecoxib has been shown to down-regulate P-gp expression. Ondansetron and fentanyl are substrates of P-gp and CNS levels are influenced by its activity. Clinically, NSAIDs augment opioid effect and reduce nausea and vomiting, possibly by preventing the CNS extrusion of opioids and ondansetron via P-gp down-regulation. We will use peripheral blood mononuclear cells P-gp activity, as measured by RT-PCR and ELISA, as a surrogate for P-gp activity at the BBB and correlate with celecoxib plasma levels. Also, there are single-nucleotide polymorphisms (SNPs) of the ABCB1 gene associated with pain and drug transport in humans (rs2032582, rs2229109, rs9282564, rs1045642 and rs1128503) and they may influence CSF drug levels including ondansetron and fentanyl based on their associated drug efflux capacity or susceptibility to celecoxib down-regulation. In addition, SNPs of the CYP2C9 P450 enzymes (rs1057910 and rs1799853) have been implicated in altered PK of celecoxib in humans. Although controversial in children, in adults they have been associated with "slow" to "poor" metabolism and increased area under the curve (AUC) up to three fold.

At our institution, children diagnosed with hematologic malignancies routinely undergo general anesthesia for bone marrow aspiration/biopsy (BM) and diagnostic/ therapeutic lumbar punctures (LP). Post intervention site pain may be associated with a post dural puncture or atypical headache. Recently there have been reports of elevated Cox-2 expression in patients with CML and lymphomas. Data suggests that the combination of Cox-2 inhibitors with standard chemotherapeutics may enhance the potential of treatment for some hematological malignancies. Access to blood and cerebral spinal fluid provide a unique opportunity to determine celecoxib concentrations in the respective compartments.

Objectives and Hypothesis:

The primary objectives are to determine CSF concentrations (ug/L) of celecoxib 121-180 minutes following ingestion of a 7 or 14 mg/kg dose of a celecoxib suspension (20 mg/ml), to develop a pediatric population-based CSF and plasma 24 hour pharmacokinetic (PK) profile of a 14 mg/kg and 7 mg/kg dose of a celecoxib suspension (20 mg/ml), and to integrate this information into a PK model that explores the relationship between plasma and CSF celecoxib concentrations and the impact of covariates using nonlinear mixed effects models.

The investigators hypothesize that a 14 mg/kg "front end loaded" dose of a celecoxib suspension (20 mg/ml) will achieve a target CSF concentration of at least 15 ug/L (equivalent to 50% of the COX-2 enzyme inhibition) approximately 121-180 minutes after oral ingestion and that these concentrations will be significantly higher than those CSF concentrations (ug/L) achieved with a 7 mg/kg traditional "allometric adjusted" dose.

Experimental Design:

This is a two-phased double-blind randomized controlled study of sixty-five (65) children aged 2-12 years in maintenance therapy for leukemia, who will receive a single dose of celecoxib prior to a scheduled lumbar puncture.

In Phase I, twenty (20) children will receive either celecoxib 14 or 7 mg/kg 121-180 minutes prior to lumbar puncture (LP). In Phase II, forty-five (45) children will receive celecoxib 14 mg/kg, 7 mg/kg or placebo in one of 5 time intervals, 1-24 hours prior to LP.

Drug levels in CSF and plasma will be measured using established HPLC-Mass Spec techniques. Pharmacogenetic data of the ABCB1 & CYP2C9 genotypes will be determined. Patient follow-up will be on Day 1 & 7 after ingestion to document adverse events.

Potential Impact:

CSF penetration of Cox-2 inhibitors may reduce the incidence of acute pain evolving into a chronic pain model. The results of this study will establish the safety of this class of medications in children and enable a more rational approach to their dosing in acute pain models and perhaps future chemotherapeutic protocols

ELIGIBILITY:
Inclusion Criteria:

Children aged 2-12 years, undergoing Maintenance phase chemotherapy for hematological malignancies and lymphomas (i.e. acute lymphoblastic leukemia [ALL] and lymphoblastic lymphomas [LLy] at CHEO. At this point, all patients would have achieved remission an average of 6 months earlier.

Exclusion Criteria:

1. Age < 2yrs and >12yrs old
2. Children with non-hematologic malignancies
3. AML
4. Children undergoing a bone marrow aspiration (BMA) only
5. Serum creatinine > 2 X UNL (upper normal limit) within 30 days
6. Abnormal liver function; alanine aminotransferase (ALT) > 2 X UNL, Aspartate aminotransferase (AST) > 2 X UNL, total & direct bilirubin > 2 X UNL within 30 days
7. History of peptic ulcer disease
8. Allergy to celecoxib or NSAIDs (note: sulpha allergy does not exclude celecoxib)
9. Recent (within 7 days) celecoxib ingestion
10. Patients receiving CYP2C9 inhibitors fluconazole, amiodarone, oxandrolone
11. Patients receiving CYP2C9 inducers rifampin and phenobarbitol
12. Patients receiving high (≥ 5 gm/m2) and/ or escalating doses of methotrexate.
13. Extremes of body mass index (BMI) (BMI <5th percentile or >95th percentile)
14. Parents of any participants, irrespective of age, who are unable to read and understand instructions relayed in English or French
15. Participant and/or parents of any participants, irrespective of age, who suffer from dementia, psychosis or any impairment that would prohibit the understanding and giving of informed consent or study-related reporting
16. Patient enrolled in another trial
17. Pregnancy.

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 65 (Estimated)
Dates: Start 2024-01-29 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Mean celecoxib CSF concentration (ug/L) within 121-180 minutes post ingestion of 7 or 14 mg/kg celecoxib. | Day 0, the day of the procedure, after taking study medication.
  Compare mean celecoxib CSF concentration (ug/L) within 121-180 minutes post ingestion of 7 or 14 mg/kg celecoxib
Mean celecoxib total and unbound plasma concentration (ug/L) in the following time intervals (mins): 0-30, 31- 60, 61- 90, 91- 120, 121-180, 181-300, 301-900 and 901-1440. | Day 0, the day of the procedure, after taking study medication.
  Compare mean celecoxib total and unbound plasma concentration (ug/L) post ingestion of 7 or 14 mg/kg celecoxib
Mean celecoxib CSF concentration (ug/L) at the following time intervals (mins): 0-60, 61-120,121-180,181-300, 301-900 and 901-1440. | Day 0, the day of the procedure, after taking study medication.
  Compare mean celecoxib CSF concentration (ug/L) post ingestion of 7 or 14 mg/kg celecoxib
Develop a PK model that explores the relationship between plasma and CSF celecoxib concentrations and the impact of covariates including age, weight and genetics using nonlinear mixed effects models. | Day 0, the day of the procedure, after taking study medication.
  The PK model will be used to see if there is a correlation between plasma and CSF celecoxib concentrations and various factors such as age, weight and genetics.

SECONDARY OUTCOMES:
Ratio CSF/unbound plasma concentration | Day 0, the day of the procedure, after taking study medication.
  Ratio CSF/unbound plasma concentration at approximately the following time intervals (mins): 0-60, 61-120,121-180,181-300, 301-900 and 901-1440.
Determine Peak Plasma concentration value (Cmax) | Day 0, the day of the procedure, after taking study medication.
  Primary outcomes 2-3 will be used to determine plasma and CSF mean +/- SD values for Maximum concentration (Cmax [ug/L])
Determine Area under the plasma concentration versus time curve (AUC) | Day 0, the day of the procedure, after taking study medication.
  Primary outcomes 2-3 will be used to determine Area under concentration curve from time 0 to infinity (AUC (0-∞) [ug/L∙h]).
Determine apparent oral volume of distribution (Vd/F [L/kg]) | Day 0, the day of the procedure, after taking study medication.
  Primary outcomes 2-3 will be used to determine apparent oral volume of distribution (Vd/F [L/kg]).
Determine apparent oral clearance (CL/F [L∙h-1∙kg-1] | Day 0, the day of the procedure, after taking study medication.
  Primary outcomes 2-3 will be used to determine apparent oral clearance (CL/F [L∙h-1∙kg-1]
Determine terminal elimination half -life (t1/2 [h]). | Day 0, the day of the procedure, after taking study medication.
  Primary outcomes 2-3 will be used to determine terminal elimination half -life (t1/2 [h]).
Determine median value for time to maximum concentration (tmax[h]). | Day 0, the day of the procedure, after taking study medication.
  Primary outcomes 2-3 will be used to determine a median value for time to maximum concentration (tmax[h]).
Pain scores versus total plasma celecoxib concentration | Day 0, the day of the procedure, after taking study medication.
  Figure depicting pain scores versus total plasma celecoxib concentration (ug/L).
Correlation with qualitative P-gp expression | Day 0, the day of the procedure, after taking study medication.
  Correlation between mononuclear cell quantitative and qualitative P-gp expression and plasma celecoxib concentrations.
Correlation between CSF and plasma study drug concentrations | Day 0, the day of the procedure, after taking study medication.
  Correlation between CSF ondansetron and fentanyl concentrations and both plasma celecoxib as well as ondansetron and fentanyl concentrations.
Pharmacogenetic data of the CYP2C9 genotypes | Day 0, the day of the procedure, after taking study medication.
  Correlation between the various P450 liver enzyme alleles encoded by the CYP2C9 gene and celecoxib plasma and analgesic concentrations.
Pharmacogenetic data of the ABCB1 genotypes | Day 0, the day of the procedure, after taking study medication.
  Correlation between various P-gp SNPs encoded by the MDR1 (ABCB1) gene and CSF fentanyl and ondansetron concentrations.
Determine study drug adverse events (AEs) | Day 0, the day of the procedure, after taking study medication.
  Compare AEs between groups and placebo within a 24 hour and 7 day period post ingestion of the study drug.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Kimmo Murto, MD, Principal Investigator — Children's Hospital of Eastern Ontario
Locations (1):
- Children's Hospital of Eastern Ontario, Ottawa, Ontario, Canada

REFERENCES:
- See also: Link to Children's Hospital of Eastern Ontario anesthesiology research page. — https://www.cheoresearch.ca/research/areas/anesthesiology/